CLINICAL TRIAL: NCT02798185
Title: Diagnostics, Imaging And Genetics Network for the Objective Study and Evaluation of Chronic Traumatic Encephalopathy (DIAGNOSE CTE) Research Project
Brief Title: The DIAGNOSE-CTE Research Project
Acronym: DIAGNOSE-CTE
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Mayo Clinic (Other); Banner Health (Other); Brigham and Women's Hospital (Other); NYU Langone Health (Other); The Cleveland Clinic (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: H-34799; U01NS093334 (NIH)
Record Dates: First submitted 2016-05-20; First posted 2016-06-14 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Chronic Traumatic Encephalopathy
MeSH Terms: conditions — Chronic Traumatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen samples to be collected include: saliva, blood and cerebral spinal fluid (CSF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Former NFL Players: 120 former National Football League players with and without reported cognitive, mood and behavior symptoms will be enrolled in this study.
- Former College Football Players: 60 former college football players with and without reported cognitive, mood and behavior symptoms will be enrolled in this study.
- Control Group: 60 asymptomatic same-age men without any history of participation in contact sports, military service, or traumatic brain injury will be enrolled in this study.

SUMMARY:
This is a study to develop methods of diagnosing chronic traumatic encephalopathy (CTE) during life, as well as to examine possible risk factors for this neurodegenerative disease. One component of this study is the use of an investigational PET scan radio tracer to detect abnormal tau protein in the brain.

DETAILED DESCRIPTION:
Chronic Traumatic Encephalopathy (CTE) is a neurodegenerative disease characterized by a distinct deposition of phosphorylated tau (p-tau) in neurons and astrocytes in a pattern that is unique from other tauopathies, including Alzheimer's disease (AD). Although the neuropathological features of CTE have become further clarified in recent years, the clinical presentation of CTE is still not well characterized. Diagnostic criteria have only recently been published and lack validation.

Neuroimaging and fluid biomarkers developed for the diagnosis of other neurodegenerative diseases have only been used in preliminary studies of individuals at high risk for CTE, namely athletes with histories of significant exposure to repetitive head impacts (RHI), such as former football players and boxers. There is thus an urgent need to develop accurate methods for detecting and diagnosing CTE during life so that effective interventions for prevention and treatment can be developed. Moreover, though a history of RHI is a necessary risk factor for CTE, it alone is not sufficient. There is a need to understand what specific aspects of RHI exposure places an individual at increased risk for CTE and to examine potential genetic polymorphisms that modify that risk.

To address these needs, the investigators are conducting a multidisciplinary, multicenter, longitudinal study of former NFL and varsity college football players (with and without symptoms), and a control group of asymptomatic same-age men without any history of RHI exposure, traumatic brain injury or military service. Subjects will be seen at 1 of 4 participating study sites in Boston; Las Vegas, ; New York; and Scottsdale/Phoenix . Subjects will undergo a baseline evaluation and a 3 year follow-up evaluation (currently former college players will not complete the follow-up evaluation). Each evaluation will be take place over a 3 day period and consist of the following procedures/tests: neurocognitive testing, determination of functional independence, neuropsychiatric examination (with measures of mood and behavior), neurological assessment (motor, headache, postural stability), neuroimaging (including structural, diffusion, functional, biochemical, and molecular imaging), lumbar punctures (for Cerebrospinal Fluid (CSF) biomarkers), blood draws (for blood biomarkers and DNA), and saliva samples (for biomarkers).

ELIGIBILITY:
Inclusion Criteria:

Former NFL Players:

* English as primary language
* No MRI or Lumbar Puncture (LP) contraindications
* Have played ≥12 years of organized football (including =>3 in college and =>3 seasons in the NFL)
* Must have played one of following positions offensive lineman, defensive lineman, linebacker, tight end, wide receiver, running back, or defensive back.
* Agree to provide name and contact information of a study partner who will complete questionnaires regarding subject's mood, behavior, thinking and cognitive function should the subject enroll in the study.

Former Collegiate Football Players

* English as primary language
* No MRI or Lumbar Puncture (LP) contraindications
* Must have played =>6 years of organized football (with => 3 years at the college level, but no organized football or other contact sport following college.)
* Must have played one of following positions offensive lineman, defensive lineman, linebacker, tight end, wide receiver, running back, or defensive back.
* No military service
* Agree to provide name and contact information of a study partner who will complete questionnaires regarding subject's mood, behavior, thinking and cognitive function should the subject enroll in the study.

Control Group

* English as primary language
* No MRI or Lumbar Puncture (LP) contraindications
* No history of organized contact sports or known traumatic brain injury (TBI) and/or moderate/severe concussions
* No history of participation in any of the following organized sports at any level: football, hockey, rugby, soccer, lacrosse, wrestling, boxing, gymnastics, martial arts, and kickboxing.
* No military service.
* Must have BMI >=24
* Must have at least 2 years post-secondary education at a 4-year accredited college or university, or have an associate's degree if they did not attend a 4-year accredited college or university
* Must have never been diagnosed with, or treated for, any of the following: depression, manic-depressive or bipolar disorder, anxiety, or other psychiatric or mental health problems
* Agree to provide name and contact information of a study partner who will complete questionnaires regarding subject's mood, behavior, thinking and cognitive function should the subject enroll in the study.
* Must be asymptomatic when screened by telephone.

Former NFL and Varsity Collegiate Football Players Exclusion Criteria:

* If they do not meet inclusion criteria
* If they have a history of clinical stroke confirmed on neuroimaging
* If they have vision or hearing impairment significant enough to compromise neuropsychological testing
* If they have been hospitalized or treated in an emergency room following a severe injury to their head since they stopped playing football
* If they are unable to undergo MRI/PET Scan
* If they have a spinal fusion at L3-4 and/or L4-5
* If they are unable to travel to one of 4 study sites to participate
* If they are an insulin dependent diabetic
* If they cannot provide the name and contact information of an eligible study partner
* If they are taking blood thinners that would make LP unsafe
* If they have a type of abnormal heart rhythm called Torsades de pointes AKA TdP
* If they have an abnormal heart rhythm disorder called QT Prolongation or take certain medications known to cause QT Prolongation
* If they do not agree to all study tests and procedures
* If they are unable to consent to study procedures

Control Group Exclusion:

* If they do not meet inclusion criteria
* If they have vision or hearing impairment significant enough to compromise neuropsychological testing
* If they are unable to undergo MRI/PET Scan
* If they have a spinal fusion at L3-4 and/or L4-5
* If they are an insulin dependent diabetic
* If they are unable to travel to one of 4 study sites to participate
* If they cannot provide the name and contact information of an eligible study partner
* If they report any cognitive concerns or dementia during screening process
* If they have a type of abnormal heart rhythm called Torsades de pointes AKA TdP
* If they have an abnormal heart rhythm disorder called QT Prolongation or take certain medications known to cause QT Prolongation
* If they are unable to consent to study procedures

Ages: 45 Years to 74 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Former National Football League Players, Former Varsity Level College Football Players, Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Neuroimaging Positron Emission Tomography for Amyloid Biomarker | One-Time
  Subjects will undergo a Florbetapir Positron Emission Tomography (PET) scan.
  The Outcome Measurement for the Florbetapir PET Scan will be "elevated" or "not elevated"
Fluid Biomarkers | 3 Years
  The following Biospecimens will be collected from subjects:
  Saliva, blood and cerebral spinal fluid (CSF). CSF will be collected by a lumbar puncture (spinal tap) Fluid biomarkers will be analyzed for the in vivo detection of CTE.
Neuropsychiatric and Neurocognitive Tests | 3 years
  Composite scores (presented as z scores) based on factor analytic methodology in the following domains:
  * Mood
  * Behavior Regulation
  * Attention, Information Processing and Psychomotor Speed
  * Executive Functioning
  * Verbal Memory
  * Visual Memory
  * Visual-Spatial Ability
  * Language
Neurological Evaluation | 3 years
  Subjects will undergo The Movement Disorder Society's Unified Parkinson's Disorders Rating Scale (MDS-UPDRS) Neurological Evaluation by a physician. This evaluation will be analyzed to characterize the clinical presentation of CTE.
Magnetic Resonance Imagining Biomarkers | 3 years
  Subjects will undergo Diffuser Tension Imaging (dti) and Functional MRI scans, to assess structural brain volumetrics, fractional anisotropy, radial diffusivity, and changes in brain activity associated with blood flow.
Neuroimaging Positron Emission Tomography for Tau Biomarker | 3 years
  Subjects will undergo an Investigational drug: AV1451 Positron Emission Tomography (PET) scan.
  The Outcome Measurement for AV1451 PET scan will be Standardized Uptake Value Ratio (SUVR) of Tau.
Magnetic Resonance Spectroscopy Biomarkers | 3 years
  Subject will also undergo Magnetic Resonance Spectroscopy (MRS) to measure glutamate, glutamine and myoinosotol.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Stern, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with FITBIR and other data sharing portals

REFERENCES:
- [Derived] Su Y, Protas H, Luo J, Chen K, Alosco ML, Adler CH, Balcer LJ, Bernick C, Au R, Banks SJ, Barr WB, Coleman MJ, Dodick DW, Katz DI, Marek KL, McClean MD, McKee AC, Mez J, Daneshvar DH, Palmisano JN, Peskind ER, Turner RW 2nd, Wethe JV, Rabinovici G, Johnson K, Tripodis Y, Cummings JL, Shenton ME, Stern RA, Reiman EM; DIAGNOSE CTE Research Project Investigators. Flortaucipir tau PET findings from former professional and college American football players in the DIAGNOSE CTE research project. Alzheimers Dement. 2024 Mar;20(3):1827-1838. doi: 10.1002/alz.13602. Epub 2023 Dec 22. PMID 38134231
- [Derived] Stern RA, Trujillo-Rodriguez D, Tripodis Y, Pulukuri SV, Alosco ML, Adler CH, Balcer LJ, Bernick C, Baucom Z, Marek KL, McClean MD, Johnson KA, McKee AC, Stein TD, Mez J, Palmisano JN, Cummings JL, Shenton ME, Reiman EM; DIAGNOSE CTE Research Project Investigators. Amyloid PET across the cognitive spectrum in former professional and college American football players: findings from the DIAGNOSE CTE Research Project. Alzheimers Res Ther. 2023 Oct 5;15(1):166. doi: 10.1186/s13195-023-01315-5. PMID 37798671
- [Derived] Alosco ML, Mariani ML, Adler CH, Balcer LJ, Bernick C, Au R, Banks SJ, Barr WB, Bouix S, Cantu RC, Coleman MJ, Dodick DW, Farrer LA, Geda YE, Katz DI, Koerte IK, Kowall NW, Lin AP, Marcus DS, Marek KL, McClean MD, McKee AC, Mez J, Palmisano JN, Peskind ER, Tripodis Y, Turner RW 2nd, Wethe JV, Cummings JL, Reiman EM, Shenton ME, Stern RA; DIAGNOSE CTE Research Project Investigators. Developing methods to detect and diagnose chronic traumatic encephalopathy during life: rationale, design, and methodology for the DIAGNOSE CTE Research Project. Alzheimers Res Ther. 2021 Aug 12;13(1):136. doi: 10.1186/s13195-021-00872-x. PMID 34384490
- See also: Study website — http://www.diagnosecte.com